CLINICAL TRIAL: NCT05779423
Title: A Phase II Study of Core Needle Biopsy and Cryoablation of an Enlarging Tumor in Patients With Advanced Melanoma Receiving Post-progression Dual Immune Checkpoint Inhibitor Therapy
Brief Title: Cryoablation+Ipilimumab+Nivolumab in Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Meghan Mooradian, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-619
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Melanoma; Skin Cancer
Keywords: Immunotherapy; Metastatic Melanoma; Resistant Metastatic Melanoma; Skin Cancer; Cryoablation
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Ipilimumab; Nivolumab; Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ipilimumab + Nivolumab + Cryoablation (Experimental): Study will be conducted in two stages:
  Stage 1: Will enroll 15 participants, and if 6 or more have clinical benefit, the study will proceed to Stage 2.
  * Baseline CT scan.
  * Cycle 1-4: Pre-determined doses of ipilimumab and nivolumab. Medications administered under direction of treating oncologist.
  * Day 2 - 14: Core Needle Biopsy followed by cryoablation between Cycle 1 - 2
  * Surveillance CT scan at weeks 8 - 12, weeks 16 - 24.
  * Follow up for 6 months to assess safety after cryoablation. Participants followed for duration of response.
  Stage 2: Will enroll 22 participants
  * Baseline CT scan.
  * Cycle 1-4: Pre-determined doses of ipilimumab and nivolumab. Medications administered under direction of treating oncologist.
  * Day 2- 14: Core Needle Biopsy followed by cryoablation between Cycle 1 - 2.
  * Surveillance CT scan at weeks 8 - 12, weeks 16 - 24
  * Follow up period to assess safety 6 months after cryoablation. Patients followed for duration of response.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Procedure: Cryoablation

INTERVENTIONS:
Drug: Ipilimumab — Monoclonal antibody administered through intravenous infusion
  Other Names: Yervoy
Drug: Nivolumab — Monoclonal antibody administered through intravenous infusion
  Other Names: Opdivo
Procedure: Cryoablation — Procedure of freezing a tumor performed via CT-guidance by interventional radiologist.

SUMMARY:
The aim of this study is to find out whether the combination of two approved drugs, ipilimumab and nivolumab, in combination with cryoablation are safe and effective for participants who have an unresectable melanoma that is resistant, or is growing, after receiving immunotherapy with a PD-1 inhibitor.

The names of the study interventions involved in this study are:

* Cryoablation (an interventional radiology procedure that freezes part of a tumor)
* Ipilimumab (an immunotherapy)
* Nivolumab (an immunotherapy)

DETAILED DESCRIPTION:
This is a single-arm, two-stage, Phase II clinical trial to test the safety and effectiveness of an investigational treatment, the combination of ipilimumab and nivolumab with cryoablation, for the treatment of metastatic melanoma resistant to PD-1 inhibition.

Ipilimumab and nivolumab are types of inhibitors. Ipilimumab targets and blocks specific proteins in cancer cells which are responsible for stopping the immune system from working correctly. Nivolumab targets a receptor on cancer cells that causes programmed cell death.

The U.S. Food and Drug Administration has approved Ipilimumab and Nivolumab for the treatment of melanoma.

Cryoablation is an approved procedure that consists of freezing a tumor and surgically removing it. The use of the study drugs and cryoablation combination is experimental.

Study procedures including screening for eligibility, study treatment including in-clinic visits, blood sample collections, Computerized Tomography (CT) scans, and tumor biopsies.

Participation in this research study is expected to last up to 3 years.

It is expected that about 37 people will take part in this research study.

The William M. Wood Foundation is supporting this research by providing funding for the cryoablation and research activities.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18) with unresectable melanoma who have progressed on immune checkpoint inhibitor therapy (pembrolizumab, nivolumab, nivolumab-relatimab, atezolizumab, ipilimumab) and for whom their treating physician plans to initiate dual ICI with ipilimumab and nivolumab. Progression on adjuvant PD-1 inhibition is permitted. PD-1 does not have to be the last therapy received. This is no limited on prior lines of ICI received. There is no wash-out period required from the time of their last therapy.
* Patients are medically eligible for dual checkpoint inhibition (i.e. no untreated/uncontrolled intercurrent medical issue including ongoing immune-related adverse event or need for systemic steroids >10mg PO prednisone or its equivalent, ECOG PS ≤2) with ipilimumab 3mg/kg and nivolumab 1mg/kg by their treating physician
* Must have a tumor amenable to percutaneous image-guided cryoablation based on routine Interventional Radiology criteria.
* Patients must have measurable disease (by RECIST) independent of the lesion to be ablated. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 (Measurement of Effect) for evaluation of measurable disease.
* Prior radiation therapy to any site is allowed; with an exception of the target site for planned cryoablation
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Life expectancy of greater than 3 months
* Participants must have adequate organ and marrow function as defined below:

  * Leukocytes ≥3,000/mcL
  * Absolute neutrophil count ≥1,000/mcL
  * Platelets ≥75,000/mcL
  * Total bilirubin ≤3 institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤5 × institutional ULN
  * CrCL > 30 ml/min
* Known Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial. (HIV testing not required at screening).
* For participants with known evidence of known chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. (HBV testing not required at screening).
* Participants with a history of known hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load. (HCV testing not required at screening).
* Participants with asymptomatic brain metastases are eligible.
* Participants with new or progressive asymptomatic brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Lesion to undergo cryoablation cannot have had prior radiation therapy or other locoregional therapy
* Inability to hold systemic anticoagulation prior to cryoablation (if holding anticoagulation is required by the operator)
* Participants who are receiving an investigational agent(s).
* Participants who are progressing on combination ipilimumab/nivolumab as their last line of therapy
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1)
* Patients with symptomatic brain metastasis or LMD
* Participants on > 10mg of oral prednisone or its equivalent
* Participants with uncontrolled intercurrent illness.
* Pregnant women are excluded from this study because immune checkpoint inhibitors have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with immune checkpoint inhibitors, breastfeeding should be discontinued.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-09-23 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Clinical Benefit | 6 months post-1st cryoablation
  Defined as the proportion of participants with best overall response per RECIST v1.1 of confirmed complete or partial response or stable disease.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | Baseline to 3 months post-cryoablation
  Defined as all adverse events (grade 1- 5) occurring during the trial and follow-up period will be summarized using CTCAE v5.0 and the Kaplan-Meier method.
Duration of Overall Response | 6 months post-1st cryoablation
  Defined as the time interval between the first declaration of response/stable disease and date of disease progression per RECIST v1.1 criteria and summarized using the Kaplan-Meier method.
Progression-Free Survival (PFS) | 6 months post-1st cryoablation
  Defined as the time interval between study enrollment and documented progression of disease per RECIST v1.1 criteria and summarized using the Kaplan-Meier method.
Overall Survival (OS) | 6 months post-1st cryoablation
  Assessed per RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan J Mooradian, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation